CLINICAL TRIAL: NCT03911934
Title: Polypharmacy Outpatient Clinic as a Randomized Intervention: Effect on Quality of Life, Admissions and Mortality
Brief Title: Polypharmacy Outpatient Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Jonatan Kornholt, MD, clinical assistent, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Polyamb-01
Record Dates: First submitted 2019-02-20; First posted 2019-04-11 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Polypharmacy
Keywords: Polypharmacy; Medication review; Randomized; Deprescribing
MeSH Terms: interventions — Medication Review; Geriatric Assessment

STUDY DESIGN:
Intervention Model Description: Randomized, parallel clinical trial with two arms. The participants are randomized to usual care or usual care plus polypharmacy intervention when they are referred to the geriatric outpatient clinic before the first visit. They stay in the assigned group until end of trial (after 13 months follow-up). Randomization is performed by the medical secretaries in the outpatient clinic in REDCap's randomization module and randomization is stratified on gender, age group (65-70 years, 71-80 years, >80 years) and number of drugs (9-11 drugs, 12-16 drugs, >16 drugs).
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor of the 13 months follow-up EQ5D data is blinded to participant allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Usual care in the geriatric outpatient clinic.
  Interventions: Other: Usual care
- Usual care plus polypharmacy intervention (Experimental): Usual care in the geriatric outpatient clinic plus polypharmacy intervention. Polypharmacy intervention consists of a medication review by a physician from the Department of Clinical Pharmacology plus additional communication with patients' GPs before and after the visit in the outpatient clinic.
  Interventions: Other: Polypharmacy intervention; Other: Usual care

INTERVENTIONS:
Other: Polypharmacy intervention — A physician from the Department of Clinical Pharmacology prepares a critial medication review before the first visit in the outpatient clinic through critical review of the patient's medical journal and communication with the patient's GP. During the visit in the outpatient clinic, medications are changed based on the medication review with consent from the patient. After the visit the GP is notified of the changes. It is possible to see the patient more than one time in the outpatient clinic (might be needed if tapering or lots of changes) and possible to follow-up on medication changes by telephone with the patient.
  Other Names: Medication review
  Arms: Usual care plus polypharmacy intervention
Other: Usual care — Usual care in the geriatric outpatient clinic with geriatric assessment from a trained geriatrician
  Other Names: Geriatric assessment

SUMMARY:
To investigate the effect of physician-initiated, medication reviews in geriatric patients on self-reported health-related quality of life, admissions, mortality and falls.

DETAILED DESCRIPTION:
Aim: To investigate the effect of physician-initiated, medication reviews in geriatric patients on self-reported health-related quality of life, admissions and mortality.

Trial design: Randomized trial with polypharmacy intervention in addition to standard geriatric care. After referral to the geriatric outpatient clinic (but before the first visit), a medical secretary screens the patient's medication on the electronic medication list. If the patient is taking more than 8 different drugs, the patient is randomized to either standard geriatric care or standard geriatric care plus polypharmacy intervention. During the first visit, the patient is informed of the project and asked for written, informed consent. If given, we collect data regarding the patient's medication and any medication changes during the intervention, demographics, frailty (FRAIL Scale), Charlson Comorbidity Index, self-reported history of falls, recent admissions, self-reported, health-related quality of life (EQ-5D-5L) and death. Data is collected at baseline, 4 months follow-up and 13 months follow-up.

Participants: All randomized, polymedicated (>8 drugs) patients referred to the geriatric outpatient clinic.

Outcomes: The primary outcome is the between-group difference in the EQ-5D-5L difference (self-reported, health-related quality of life) between baseline and 13 month follow-up.

The secondary outcomes are number of medications, number of successful medication discontinuations, number of admissions and visits to the emergency department, self-reported low-energy falls, and death.

ELIGIBILITY:
Inclusion Criteria:

* New referral to the geriatric outpatient clinic
* More than > 8 different substances in drugs on the electronic medication list before the first visit. Regular and PRN drugs count. Excluding topical treatment (eye drops, ear drops, creams etc) but including inhalation, excluding antibiotics with limited duration, excluding multivitamins, and excluding protein drinks.

Exclusion Criteria:

* Inability (or refuses) to give informed consent (e.g. because of lack of interest, inability to understand the intervention or language barriers).
* Inability to understand the consent form and/or the intervention.
* Patients referred to the dementia diagnostics unit.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 408 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
EQ5D-5L index, 4 months, including death | EQ5D-5L index values at baseline (inclusion) and at 4 months followup
  Comparison of changes in EQ5D-5L index from baseline to 4 months follow-up between the control and intervention group (including death). EQ-5D is an abbreviation for "European Quality of life - 5 Dimensions" and measures Quality of Life. The scale has five subcomponents with scores from 1 (best) to 5 (worst). The five subcomponents consitute a health state that is translated into an index value using the Danish EQ-5D-5L Value Set from 2021 (see Jensen et al. The Danish EQ-5D-5L Value Set: A Hybrid Model Using cTTO and DCE Data. Appl Health Econ Health Policy. 2021 Feb 2. doi: 10.1007/s40258-021-00639-3. PMID: 33527304). The index value is anchored at 0 = death and 1 = full health and the range in the Danish population ranges from -0.758 (worse than death) to 1.0 (full health). Higher values / increases in index value is better than lower values / decreases in index value.

SECONDARY OUTCOMES:
EQ5D-5L index, 13 months, including death | EQ5D-5L index values at baseline (inclusion) and at 13 months follow-up
  Comparison of changes in EQ5D-5L index from baseline to 13 months follow-up between the control and intervention group (including death). EQ-5D is an abbreviation for "European Quality of life - 5 Dimensions" and measures Quality of Life. The scale has five subcomponents with scores from 1 (best) to 5 (worst). The five subcomponents consitute a health state that is translated into an index value using the Danish EQ-5D-5L Value Set from 2021 (see Jensen et al. The Danish EQ-5D-5L Value Set: A Hybrid Model Using cTTO and DCE Data. Appl Health Econ Health Policy. 2021 Feb 2. doi: 10.1007/s40258-021-00639-3. PMID: 33527304). The index value is anchored at 0 = death and 1 = full health and the range in the Danish population ranges from -0.758 (worse than death) to 1.0 (full health). Higher values / increases in index value is better than lower values / decreases in index value.
Mortality | Baseline to 13 months follow-up.
  Comparison of time to death during the 13 month follow-up between the control and intervention group.
Admissions (number) | From baseline to 4 month follow-up and from 4 month follow-up to 13 month-followup comparison between the control and intervention group.
  Number of admissions (any cause)
Admissions (days) | From baseline to 4 month follow-up and from 4 month follow-up to 13 month-followup comparison between the control and intervention group.
  Number of admission days (any cause)
Number of drugs | At 4 month follow-up and 13 month follow-up.
  Number of prescription drugs. Comparison between the control and intervention group.
Falls | Comparison between groups at 4 month follow-up and 13 month follow-up.
  Binary: Any falls the last 3 months?
EQ5D-5L index, 4 months, excluding death | EQ5D-5L index values at baseline (inclusion) and at 4 months followup
  Comparison of changes in EQ5D-5L index from baseline to 4 months follow-up between the control and intervention group (excluding death). EQ-5D is an abbreviation for "European Quality of life - 5 Dimensions" and measures Quality of Life. The scale has five subcomponents with scores from 1 (best) to 5 (worst). The five subcomponents consitute a health state that is translated into an index value using the Danish EQ-5D-5L Value Set from 2021 (see Jensen et al. The Danish EQ-5D-5L Value Set: A Hybrid Model Using cTTO and DCE Data. Appl Health Econ Health Policy. 2021 Feb 2. doi: 10.1007/s40258-021-00639-3. PMID: 33527304). The index value is anchored at 0 = death and 1 = full health and the range in the Danish population ranges from -0.758 (worse than death) to 1.0 (full health). Higher values / increases in index value is better than lower values / decreases in index value.
EQ5D-5L index, 13 months, excluding death | EQ5D-5L index values at baseline (inclusion) and at 13 months followup
  Comparison of changes in EQ5D-5L index from baseline to 13 months follow-up between the control and intervention group (excluding death). EQ-5D is an abbreviation for "European Quality of life - 5 Dimensions" and measures Quality of Life. The scale has five subcomponents with scores from 1 (best) to 5 (worst). The five subcomponents consitute a health state that is translated into an index value using the Danish EQ-5D-5L Value Set from 2021 (see Jensen et al. The Danish EQ-5D-5L Value Set: A Hybrid Model Using cTTO and DCE Data. Appl Health Econ Health Policy. 2021 Feb 2. doi: 10.1007/s40258-021-00639-3. PMID: 33527304). The index value is anchored at 0 = death and 1 = full health and the range in the Danish population ranges from -0.758 (worse than death) to 1.0 (full health). Higher values / increases in index value is better than lower values / decreases in index value.
EQ5D-5L VAS, 13 months, including death | EQ5D-5L VAS values at baseline (inclusion) and at 13 months followup
  Comparison of changes in EQ5D-5L VAS from baseline to 13 months follow-up between the control and intervention group (including death). EQ-5D is an abbreviation for "European Quality of life - 5 Dimensions" and measures Quality of Life. The visual analog scale's (VAS) range is from 0 (worst health imaginable) to 100 (best health imaginable) and the participants score their own health. Higher values / increases in EQ-5D VAS is better compared with lower values / decreases in EQ-5D VAS.
EQ5D-5L VAS, 4 months, including death | EQ5D-5L VAS values at baseline (inclusion) and at 4 months followup
  Comparison of changes in EQ5D-5L VAS from baseline to 4 months follow-up between the control and intervention group (including death). EQ-5D is an abbreviation for "European Quality of life - 5 Dimensions" and measures Quality of Life. The visual analog scale's (VAS) range is from 0 (worst health imaginable) to 100 (best health imaginable) and the participants score their own health. Higher values / increases in EQ-5D VAS is better compared with lower values / decreases in EQ-5D VAS.
EQ5D-5L VAS, 13 months, excluding death | EQ5D-5L VAS values at baseline (inclusion) and at 13 months followup
  Comparison of changes in EQ5D-5L VAS from baseline to 13 months follow-up between the control and intervention group (excluding death). EQ-5D is an abbreviation for "European Quality of life - 5 Dimensions" and measures Quality of Life. The visual analog scale's (VAS) range is from 0 (worst health imaginable) to 100 (best health imaginable) and the participants score their own health. Higher values / increases in EQ-5D VAS is better compared with lower values / decreases in EQ-5D VAS.
EQ5D-5L VAS, 4 months, excluding death | EQ5D-5L VAS values at baseline (inclusion) and at 4 months followup
  Comparison of changes in EQ5D-5L VAS from baseline to 4 months follow-up between the control and intervention group (excluding death). EQ-5D is an abbreviation for "European Quality of life - 5 Dimensions" and measures Quality of Life. The visual analog scale's (VAS) range is from 0 (worst health imaginable) to 100 (best health imaginable) and the participants score their own health. Higher values / increases in EQ-5D VAS is better compared with lower values / decreases in EQ-5D VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel B Christensen, MD, PhD, Principal Investigator — University Hospital Bispebjerg and Frederiksberg
Locations (1):
- Geriatric Outpatient Clinic, Frederiksberg Hospital, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kornholt J, Feizi ST, Hansen AS, Laursen JT, Johansson KS, Reuther LO, Petersen TS, Pressel E, Christensen MB. Medication changes implemented during medication reviews and factors related to deprescribing: Posthoc analyses of a randomized clinical trial in geriatric outpatients with polypharmacy. Br J Clin Pharmacol. 2023 Nov;89(11):3291-3301. doi: 10.1111/bcp.15805. Epub 2023 Jul 6. PMID 37254818